CLINICAL TRIAL: NCT03816826
Title: "THE EFFECTS OF LOW LEVEL LASER THERAPY VERSUS STRAIN/COUNTER STRAIN TECHNIQUE IN ACUTE SOFT TISSUE INJURIES"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Isra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1609MPHILSMMPT002
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hamstring Injury; Strain Counter Strain
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 60 athletes with hamstring injury distributed randomly into 3 group
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- laser (Experimental): athletes with acute soft tissue injuries will be recruited in the study , patients will be treated using the the laser therapy
  Interventions: Other: physical therapy
- strain/counter strain (Experimental): athletes with acute soft tissue injuries will be treated with with strain counter strain technique
  Interventions: Other: physical therapy
- combination therapy (Experimental): combination of laser therapy along with strain counter strain technique to visualize the effect the
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: physical therapy — both are physical therapy intervention technique used to treat the soft tissue acute injuries

SUMMARY:
Muscle strain injuries are common in sports but are often misdiagnosed and maltreated.

Their significance is often underestimated because most athletes can continue their daily activities soon after the injury. Proximal hamstrings strains have attracted greater attention because they have a high incidence which is approximately 42%.

DETAILED DESCRIPTION:
it will be randomized control trial with 60 patients with Acute hamstring Injuries divided into 3 groups. One group will be given Laser therapy, 2nd will be given Strain/Counter Strain technique and 3rd will be given both the techniques in combination This study will be conducted in Rehabilitation setup of Pakistan Hockey Federation Lahore, and Institute of Orthopedics and Rehabilitation Center Garden Town Lahore. Non probability Convenience Sampling technique will be utilized

ELIGIBILITY:
Inclusion Criteria:

hamstring injury patient with grade 2 or 1 both male and female local tenderness on palpation pain with resisted knee flexion pain with resisted hip extension pain on stretching of effected area

Exclusion Criteria:

* patient with fracture
* patient with grade 3 orthopedic condition like ankylosing spondylitis medically unstable

Ages: 16 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 5 days
  to measure pain scale will be used consisting of digits from 0 to 10
FASH questionaire | 5 days
  hamstring injury and funtional capacity of hamstring

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Adnan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No